CLINICAL TRIAL: NCT06956794
Title: Multimodal Training With Immersive VIRTUAL Reality to Improve the Cognitive Health and Emotional Well-being of Older Women Living Alone (VirtualDONA)
Brief Title: Multimodal Training With Immersive Virtual Reality to Improve the Cognitive Health and Emotional Well-being of Older Women Living Alone
Acronym: VirtualDONA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Broomx Technologies (Unknown); SUARA Cooperativa (Unknown)
Responsible Party: Principal Investigator, Maite Garolera, Chief of the Neuropsychological Unit and Director of the Brain, Cognition, and Behavior Research Group, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024PROD00053
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Social Isolation in Older Adults; Poverty
Keywords: Social Isolation; Cognitive Dysfunction; Aging; Poverty; Virtual Immersive Reality
MeSH Terms: conditions — Social Isolation; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two parallel groups: one receiving a multimodal group-based intervention using immersive virtual reality, and a control group maintaining usual activities. The intervention consists of 16 sessions over 8 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive VR-Based Multimodal Intervention (Experimental): Participants in this arm will receive a multimodal, group-based intervention using immersive virtual reality without headsets. The intervention includes mindfulness, cognitive training, and physical exercises delivered in 16 group sessions over 8 weeks.
  Interventions: Behavioral: VirtualDONA Multimodal Program
- Usual Activity (Control Group) (No Intervention): Participants in this arm will continue their usual daily routines with no specific intervention during the study period.

INTERVENTIONS:
Behavioral: VirtualDONA Multimodal Program — A group-based behavioral intervention using immersive virtual reality without headsets. The 8-week program includes 16 sessions combining mindfulness, cognitive training, and physical exercises, designed to improve cognitive health and emotional well-being in older women living alone and at risk of poverty.
  Arms: Immersive VR-Based Multimodal Intervention

SUMMARY:
This study aims to evaluate the effectiveness of an immersive virtual reality-based multimodal intervention (VirtualDONA) to improve cognitive health and emotional well-being in older women living alone and at risk of poverty. The intervention combines mindfulness, cognitive, and physical training in a group format over 8 weeks.

DETAILED DESCRIPTION:
The VirtualDONA project aims to promote the health of older women living alone and at risk of poverty, as they are considered a highly vulnerable population. Women's longer life expectancy compared to men leads to a greater proportion of women living alone. In Catalonia, there are 786,000 people living alone, and 42.2% are aged 65 or older. The combination of being a woman, of advanced age, and living alone is associated with a high rate of poverty.

These social and economic determinants significantly increase the likelihood of developing dementia and/or mental health disorders in affected individuals. Research has established a connection between social isolation, aging, and a higher probability of experiencing dementia, stress, depression, and anxiety. Economic uncertainty is also known to contribute to stress and anxiety, while social stigma-particularly affecting older women-can negatively impact their cognitive and mental health.

All of these factors highlight the need for preventive interventions targeting women over the age of 65 who live alone and have incomes below the minimum income threshold. VirtualDONA proposes a preventive intervention for this population using immersive virtual reality technology (without headsets) to improve cognitive functioning, emotional well-being, and quality of life.

The intervention will be delivered in a group format over 8 weeks (16 sessions). The combination of mindfulness, cognitive, and physical exercises within a virtual environment offers a suitable multimodal platform for a comprehensive and innovative intervention aimed at vulnerable women. The project aims to demonstrate the benefits of this approach and to develop a sustainable, scalable, and long-term viable business model.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 65 years or older
* Living alone
* Registered with the elderly care services of Suara Cooperativa
* Annual income below the guaranteed minimum income threshold (below €20,353.62/year)
* Global cognitive functioning not suggestive of dementia, defined as MMSE score ≥ 24
* Able to read and write
* Good command of Catalan and/or Spanish
* Signed informed consent to participate in the study

Exclusion Criteria:

* History of severe neurological, psychiatric disorders, or intellectual disability
* Uncorrected sensory deficits (e.g., vision or hearing)
* Physical or motor impairments that may interfere with participation or bias outcome measures

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in scores of global cognition | Baseline and after the 8-week intervention
  Global cognition is assessed with the Mini-Mental State Examination (MMSE), a brief screening tool for cognitive impairment. The MMSE includes items that evaluate orientation, registration, attention and calculation, recall, language, and visuospatial ability. Scores range from 0 to 30, with higher scores indicating better cognitive function.
Differences between groups in scores of global cognition | Baseline and after the 8-week intervention
  Global cognition is assessed with the Montreal Cognitive Assessment (MoCA) a screening tool designed to identify mild cognitive impairment (MCI) and other cognitive deficits. The MoCA takes around 10-15 minutes to complete and consists of 30 items (range=0-30). Higher scores mean a better outcome.
Differences between groups in scores of verbal episodic memory | Baseline and after the 8-week intervention
  Verbal episodic memory is assessed with the Free and Cued Selective Reminding Test (FCSRT), which evaluates the ability to learn and recall words with both free and cued recall conditions. The total score ranges from 0 to 48, based on the number of words correctly recalled. Higher scores indicate better memory performance.
Differences between groups in scores of auditory attention | Baseline and after the 8-week intervention
  Auditory attention is measured with Digit Span Forward from WAIS-IV. Participants are asked to repeat numbers in the same order as read aloud by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of working memory | Baseline and after the 8-week intervention
  Working memory is measured with Digit Span Backward from WAIS-IV. Participants are asked to repeat the numbers in the reverse order of that presented by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of processing speed | Baseline and after the 8-week intervention
  Processing speed is measured with the Digit Symbol Coding subtest from the WAIS-III. It consists of replacing symbols that lack verbal meaning with numbers based on a key. Higher scores indicate better outcomes.
Differences between groups in scores of visual scanning and processing speed | Baseline and after the 8-week intervention
  Visual scanning and processing speed are measured with the Trail-Making Test-A version. Participants are asked to connect a series of numbered circles on a page in numerical order. Higher scores mean a better outcome.
Differences between groups in scores of executive functioning and cognitive flexibility | Baseline and after the 8-week intervention
  Executive functioning and cognitive flexibility are measured with the Trail-Making Test-B version. Participants are asked to connect a series of circles that contain both numbers and letters in alternating numerical and alphabetical order. Higher scores mean a better outcome.
Differences between groups in scores of executive functioning | Baseline and after the 8-week intervention
  Executive functioning is assessed with the Modified Wisconsin Card Sorting Test (M-WCST), which evaluates abstract reasoning, cognitive flexibility, and the ability to shift problem-solving strategies. Performance is scored based on the number of categories completed, total errors, and perseverative errors. Higher scores in perseverative errors indicate worse performance, while more categories completed reflect better executive functioning.
Differences between groups in scores of selective attention, inhibition, and processing speed | Baseline and after the 8-week intervention
  Selective attention, inhibition, and processing speed are measured with the Stroop Color and Word Test. Participants are asked to name the color of a series of color patches (Stroop Color Naming), read a series of color words (Stroop Word Reading), and name the color of a series of color words where the word and color do not match (e.g., the word "red" written in blue ink), Stroop Color-Word Interference. Higher scores mean a better outcome.
Differences between groups in scores of phonetic fluency | Baseline and after the 8-week intervention
  Phonemic verbal fluency is assessed using the PMR test, in which participants are asked to produce as many words as possible beginning with the letters P, M, and R, one minute per letter. The total score is the sum of all correct, non-repeated words across the three trials. Higher scores indicate better phonemic fluency and executive function.
Differences between groups in scores of semantic verbal fluency | Baseline and after the 8-week intervention
  Semantic verbal fluency is assessed with a category fluency task in which participants are asked to name as many words as possible belonging to a specific semantic category (e.g., animals, fruits) within one minute. The total score is the number of correct, non-repeated words produced. Higher scores indicate better semantic fluency and lexical access.
Differences between groups in language | Baseline and after the 8-week intervention
  Language function is assessed using the 15-item version of the Boston Naming Test (BNT), a confrontation naming task consisting of 15 black-and-white line drawings of objects with increasing difficulty. The total score is the number of correctly named items. Higher scores indicate better naming ability.

SECONDARY OUTCOMES:
Differences between groups in scores of Quality of Life | Baseline and after the 8-week intervention
  Quality of Life is measured with EuroQoL-5D (EQ-5D) a self-completion questionnaire, which consists of five questions: covering mobility, hygiene, activities, pain, and anxiety. The descriptive system divides each of the 5 dimensions into three levels of response: the absence of a problem, some problem, and extreme problem. Lower scores indicate better outcomes. In addition, the questionnaire has a plus scale where the participants rated their health state on a scale of 0-100. In this scale, higher scores indicate better outcome.
Differences between groups in scores of loneliness | Baseline and after the 8-week intervention
  Loneliness levels are measured through the UCLA Loneliness Scale, a widely recognized tool for measuring subjective feelings of loneliness or social isolation. The most recent version, contains 20 items rated on a scale from 1 (Never) to 4 (Always). Higher scores indicate worse outcomes.
Differences between groups in scores of perceived social support | Baseline and after the 8-week intervention
  Perceived social support is measured with the Oslo 3-Item Social Support Scale (OSLO-3). The OSLO-3 is a brief measure of perceived social support, consisting of three items assessing the number of close confidants, perceived concern from others, and ease of obtaining practical help. Scores range from 3 to 14, with higher scores indicating greater perceived social support.
Differences between groups in scores of emotional well-being | Baseline and after the 8-week intervention
  Emotional well-being is measured with the WHO-Five Wellbeing Index Scale (WHO-5). The WHO-5 is a brief self-reported measure of current mental well-being, consisting of five positively worded items. Each item is rated on a 6-point Likert scale, resulting in a raw score ranging from 0 to 25. The score is multiplied by 4 to yield a final score ranging from 0 to 100, where higher scores indicate better well-being.
Differences between groups in scores of depression | Baseline and after the 8-week intervention
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Higher scores mean a worse outcome.
Differences between groups in scores of anxiety | Baseline and after the 8-week intervention
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in scores of frailty | Baseline and after the 8-week intervention
  Frailty is measured with the FRAIL scale. The FRAIL Scale is a 5-item screening tool that assesses frailty based on fatigue, resistance, ambulation, illnesses, and loss of weight. Each item is scored as 0 (no) or 1 (yes), with total scores ranging from 0 to 5. Higher scores indicate greater levels of frailty.
Differences between groups in scores of dietary habits | Baseline and after the 8-week intervention
  Dietary haabits are measured with the PREDIMED questionnaire (adherence to the Mediterranean diet). The PREDIMED is a 14-item questionnaire used to assess adherence to the Mediterranean diet. Each item is scored 0 or 1 depending on dietary habits, resulting in a total score ranging from 0 to 14. Higher scores indicate greater adherence to the Mediterranean diet.
Differences between groups in scores of performed physical activity | Baseline and after the 8-week intervention
  Performed physical activity is measured with The International Physical Activity Questionnaire (IPAQ) is a questionnaire composed of 7 questionsin order to assessthe frequency, duration, and intensity (vigorous or moderate) of the performed physical activity, walking, and sitting time during a business day for the last 7 days. Later, from the minutes obtained from the participant's answers, the METS (metabolic equivalent tasks) conversion is performed, allowing a classification, depending on the energy consumption obtained for each activity, into three categories (low, medium, high). Higher score indicate better outcome.
Differences between groups in scores of Sleep Quality | Baseline and after the 8-week intervention
  Sleep Quality is measured with The Pittsburgh Sleep Quality Index (PSQI). This test presents 24 items, although only 19 are taken into account for the correction. This test is divided into 7 dimensions, namely, sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, hypnotic drugs, and daytime dysfunction. Higher scores indicate worse sleep quality.

OTHER OUTCOMES:
Qualitative user experience | Within one week after the end of the 8-week intervention
  Post-intervention focus groups will explore participants' perceived cognitive and emotional benefits, program satisfaction, and usability of the immersive VR platform. Transcripts will be analyzed using thematic content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Maite Garolera, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (2):
- Spain (2):
  - SUARA Cooperativa, Barcelona, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: No